CLINICAL TRIAL: NCT00111293
Title: Top-Down Attentional Control of Visual Processing
Brief Title: Attention and Visual Perception
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050157; 05-M-0157
Record Dates: First submitted 2005-05-18; First posted 2005-05-19 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-05-14

CONDITIONS: Focal Lesions; Focal Brain Lesion
Keywords: Attention; Executive Function; Vision; fMRI; Top-Down; Visual Processing; Lesion; Prefrontal; Parietal; Focal Brain Lesion; Healthy Volunteer

SUMMARY:
The NIMH is conducting studies aimed at gaining a better understanding of the areas of the brain that are involved in different types of mental processes. This study will focus on brain regions involved in visual perception and attention.

Healthy normal volunteers and people who have had a stroke or undergone neurosurgery may be eligible for this study. Candidates must be 18 years of age or older, They must not have a history of a psychiatric disorder, including depression, anxiety, psychosis, or neurological disease other than stroke or the previous neurosurgery.

Participants undergo the following tests and procedures during four or more visits to the NIH Clinical Center:

* Physical and neurological examinations and depression rating scale.
* Cognitive testing: Subjects complete written tests, sit at a computer and make decisions about what they are shown by pressing keys, or answer questions from a test examiner.
* Behavioral training: Subjects practice performing a cognitive task that involves looking at and making decisions about visual images that appear on a computer screen.
* Magnetic resonance imaging (MRI): Subjects undergo MRI scanning while they perform the task they previously practiced. The MRI scanner is a metal cylinder surrounded by a strong magnetic field. During the procedure, subjects lie still for up to 10 minutes at a time on a table that can slide in and out of the cylinder. The entire MRI scanning session takes about one hour. There are multiple scans which each can take up to 10 minutes. They may be asked to return for one or two additional scanning sessions.

During the behavioral training or MRI scanning, special pieces of equipment that monitor eye movements may be used.

Some subjects may be asked to return to NIH for an additional visit to participate in a magnetoencephalographic scan. This test uses several sensors applied to the scalp to measure very small changes in magnetic fields. This is another way to measure brain activity.

DETAILED DESCRIPTION:
Attention is required for most, if not all, perceptual processes. There is a converging body of evidence from single-cell recording studies in monkeys and neuroimaging, behavioral, and clinical studies in humans showing that the processing of attended information is enhanced relative to the processing of unattended information.

What is the source of this attentional modulation? Because neuroimaging studies have demonstrated that multiple cortical regions are recruited during tasks involving selective attention, it has proven difficult thus far to determine the differential contributions of each region. A central goal of the proposed research is to characterize the contributions of prefrontal cortex and parietal cortex and test the hypothesis that these regions exert top-down modulatory influences over visual processing areas. Specifically, we wish to investigate the interaction between areas involved in attentional control and visual areas modulated by attention.

We propose to study patients with focal lesions and normal volunteers while they perform tasks requiring attention. Subjects will participate, first, in a series of behavioral studies involving selective attention; the relative performance of different patient groups and neurologically normal volunteers will be compared. Subjects will also be studied while performing similar tasks during functional magnetic resonance imaging (fMRI). We hypothesize that selective attention will be heavily impaired by lesions of key prefrontal (e.g., dorsolateral prefrontal cortex) and key parietal (e.g., superior parietal lobule) sites. We also expect that brain imaging data will show decreased activation in visual regions ipsilateral to the focal lesions in prefrontal and parietal cortex, thus providing evidence that prefrontal and parietal cortex are sources of top-down modulation. Although other research groups have compared the behavior of patients with various focal lesions or have performed fMRI studies of visual attention in neurologically normal patients, we are unaware of any concerted effort to perform fMRI in patients with focal lesions in order to functionally isolate the contributions of individual cortical regions that serve as critical nodes in the attentional network.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALL SUBJECTS -

All subjects will be volunteers and be 18 years of age or older.

PATIENTS -

Subjects with unilateral or bilateral lesions of prefrontal or parietal cortex will be selected for participation in the behavioral and brain-imaging studies described within this protocol.

Control subjects with unilateral or bilateral lesions of temporal cortex will also be studied.

Finally, patients with amygdala lesions will also be studied to test the specific hypothesis outlined in Experiment 4.

In order to obtain a sufficient number of focal lesion patients representative of different brain regions, patients with different etiologies will be studied, provided the damage is circumscribed.

The main etiologies that we will consider are stroke, lobectomy, and tumor.

We will restrict groups to include patients with the same etiology, lesion location, and lesion volume. Lesion location will consider the two hemispheres separately.

Patients who also have non-amygdala subcortical lesions will be grouped separately from patients with cortical-only lesions.

Our goal is to not group patients with more focal brain lesions compromising a single region (e.g., middle frontal gyrus) with patients with more massive damage (e.g., large extents of superior, middle, and inferior frontal gyrus).

Focal lesion patients will not be excluded on the basis of medication.

NORMAL VOLUNTEERS -

Neurologically normal, age-matched volunteers will be recruited from the local community through normal Clinical Center channels.

EXCLUSION CRITERIA:

The following criteria will be used to exclude patients or healthy volunteers from participation in this study:

* Patients with language impairments that prevent them from understanding our tasks or follow instructions will be excluded.
* Patients with a WAIS-R Full-Scale IQ of less than 75 will be excluded.
* Patients with severe cognitive dysfunction as assessed by the neuropsychological tests.
* Subjects with moderate or severe depression as assessed by the Beck Depression Inventory (scores greater than 18).
* Patients who cannot perform control tasks to the same level of performance as the control subjects will be excluded.
* Subjects with contraindication to MRI scanning will be excluded from any testing which involves the use of MRI. These contraindications include subjects with the following devices or conditions: a) central nervous system aneurysm clips; b) implanted neural stimulator; c) implanted cardiac pacemaker or defibrillator; d) cochlear implant; e) ocular foreign body (e.g., metal shavings); f) insulin pump; g) metal shrapnel or bullet; h) any implanted device that is incompatible with MRI.
* Subjects with a history of any neurological or psychiatric disorder not related to the focal lesion (e.g., epilepsy, schizophrenia, etc.)
* Subjects with any previous head injuries not related to the focal lesion.
* Subjects with a history of drug or alcohol abuse or addiction (determined by a qualified neurologist/psychiatrist).
* Subjects with conditions that preclude entry into the scanner (e.g., morbid obesity, claustrophobia, etc.) will not be included in brain imaging studies.
* Female subjects of child-bearing age will be excluded from brain imaging studies if they are pregnant or refuse to undergo a urine pregnancy test.
* Subjects with visual, auditory, motor, or language problems that would prohibit them from being able to properly perform the visual attention tasks, to understand instructions, indicate their responses, or to communicate with the experimenter via an intercom system.
* Subjects who have undergone radiation treatment or chemotherapy during a one-year period prior to the experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-05-16; Study Completion 2010-05-14

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anderson AK, Phelps EA. Lesions of the human amygdala impair enhanced perception of emotionally salient events. Nature. 2001 May 17;411(6835):305-9. doi: 10.1038/35077083. PMID 11357132
- [Background] Barcelo F, Suwazono S, Knight RT. Prefrontal modulation of visual processing in humans. Nat Neurosci. 2000 Apr;3(4):399-403. doi: 10.1038/73975. PMID 10725931
- [Background] Bechara A, Damasio H, Damasio AR. Emotion, decision making and the orbitofrontal cortex. Cereb Cortex. 2000 Mar;10(3):295-307. doi: 10.1093/cercor/10.3.295. PMID 10731224